CLINICAL TRIAL: NCT07150260
Title: Evaluation of the Correlation Between Carotid Stump Pressure and Interhemispheric rSO₂ Asymmetry in Awake Carotid Endarterectomy: A Prospective Cohort Study
Brief Title: Correlation Between Carotid Stump Pressure and Interhemispheric rSO₂ Asymmetry During Awake Carotid Endarterectomy
Status: Recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ahmet Salih Tüzen, MD, Principal Investigator, Department of Anesthesiology and Reanimation, Izmir Katip Celebi University
Other Study IDs: 2025-0442
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Carotid Artery Stenosis Symptomatic; Carotid Endarterectomy (CEA) Surgical Patients; Cerebral Hypoperfusion
Keywords: Carotid stump pressure; Near-infrared spectroscopy; rSO₂ asymmetry; Cerebral oxygenation; Awake carotid endarterectomy; Regional anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Asymmetry Group (>10% rSO₂ Difference): This group includes patients who exhibit a significant interhemispheric cerebral oxygenation asymmetry during awake carotid endarterectomy, defined as an absolute difference in ΔrSO₂ greater than 10% between the ipsilateral (surgical) and contralateral hemispheres.
- Cerebral Symmetry Group (≤10% rSO₂ Difference): This group includes patients who exhibit a nonsignificant interhemispheric cerebral oxygenation asymmetry during awake carotid endarterectomy, defined as an absolute difference in ΔrSO₂ lesser than 10% between the ipsilateral (surgical) and contralateral hemispheres.

SUMMARY:
This study aims to better understand how well the brain is perfused (supplied with blood and oxygen) during a specific type of surgery called carotid endarterectomy (CEA), which is performed to prevent strokes in people with stenosis of carotid arteries.

During this surgery, the surgeon temporarily clamps the carotid artery to remove a blockage, which can reduce blood flow to the brain. Monitoring brain oxygen levels during this time is important to prevent brain injury. Two common monitoring methods are:

Stump pressure (SP) - a pressure measurement taken from the carotid artery during surgery.

Near-infrared spectroscopy (NIRS) - a non-invasive technique that tracks brain oxygen levels in real time.

This study focuses on the relationship between carotid stump pressure and differences in brain oxygenation between the two sides of the brain (interhemispheric asymmetry), as measured by NIRS.

The study will include patients undergoing awake CEA (under regional anesthesia) at a single center university hospital. Oxygen levels in both hemispheres of the brain will be monitored before and after the carotid artery is clamped after 3 minutes. Stump pressure will also be measured. The researchers will examine whether low stump pressure is linked to greater differences in brain oxygen levels between the two sides.

The primary goal is to determine whether a large difference in brain oxygenation between the two hemispheres (greater than 10%) is associated with low carotid stump pressure. Secondary goals include identifying a stump pressure threshold that predicts significant asymmetry and analyzing the influence of patient and surgical factors.

The findings may help improve how surgeons and anesthesiologists monitor and protect the brain during CEA, particularly in patients who are awake and can be observed for neurological changes.

DETAILED DESCRIPTION:
Carotid artery stenosis accounts for approximately 15-30% of ischemic strokes, highlighting the importance of carotid endarterectomy (CEA) as a preventive surgical strategy. One of the most critical intraoperative concerns during CEA is cerebral hypoperfusion at the time of carotid cross-clamping, when antegrade ipsilateral blood flow is interrupted. Monitoring cerebral oxygenation and collateral circulation during this period is essential to reduce the risk of ischemic complications. Traditionally, carotid stump pressure (SP) measurement has been used as a surrogate of collateral flow, whereas near-infrared spectroscopy (NIRS) provides a continuous, non-invasive estimate of regional cerebral oxygen saturation (rSO₂). While both tools are widely used, each has limitations, and there is no universal consensus on their predictive thresholds. Recent interest has shifted toward analyzing interhemispheric asymmetry in rSO₂ as a potentially physiological marker of cerebral perfusion adequacy in other clinical conditions.

This prospective, single-center observational cohort study will evaluate the association between carotid stump pressure and interhemispheric rSO₂ asymmetry in patients undergoing awake CEA under regional anesthesia. All patients will undergo awake CEA under regional anesthesia (superficial cervical plexus block) with bilateral NIRS monitoring and intraoperative stump pressure measurement. Data will be collected at baseline (before cross-clamping) and 3 minutes after carotid cross-clamp application. Patients will be stratified into two groups based on interhemispheric ΔrSO₂ asymmetry (>10% vs. ≤10%).

The primary objective is to determine whether stump pressure values differ significantly between patients with interhemispheric rSO₂ asymmetry greater than 10% (asymmetry group) compared with those with asymmetry of 10% or less (symmetry group).

Secondary objectives include:

Interhemispheric asymmetry difference;

Assessing the correlation between SP and interhemispheric ΔrSO₂ difference;

Assessing the correlation between SP and ipsilateral ΔrSO₂;

Identifying a carotid SP threshold predictive of significant interhemispheric asymmetry using receiver operating characteristic (ROC) curve analysis;

Evaluating the independent predictive value of SP for cerebral asymmetry using multivariable logistic regression adjusted for age, sex, degree of carotid stenosis, and intraoperative hemodynamic variables;

Comparing intraoperative hemodynamic parameters (PaO₂ (partial pressure of arterial oxygen), SpO₂ (peripheric oxygen saturation), systolic blood pressure, and heart rate) and procedural variables (need for shunt, cross-clamp duration, surgical time) between groups;

Documenting postoperative complications, including neurological deficits or bleeding, within 30 days of surgery.

A power analysis based on preliminary data (SP = 56 ± 15 mmHg in the symmetry group vs. 44 ±13 mmHg in the asymmetry group) yielded an effect size (Cohen's d) of 0.855. With α = 0.05 and 90% power, a minimum of 30 patients per group (60 total) are required to detect a significant difference in stump pressure between groups.

The findings of this study may refine intraoperative brain monitoring practices during CEA by clarifying the physiological relationship between stump pressure and cerebral oxygenation asymmetry.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for elective carotid endarterectomy (CEA)
* Able to tolerate surgery under regional anesthesia (superficial cervical plexus block)
* Availability of bilateral regional cerebral oxygen saturation (rSO₂) measurements by near-infrared spectroscopy (NIRS)
* Successful intraoperative carotid stump pressure (SP) measurement after cross-clamping
* Provided written informed consent

Exclusion Criteria:

* Incomplete NIRS or SP recordings
* Conversion from regional to general anesthesia
* Intraoperative technical complications preventing monitoring
* History of prior ipsilateral carotid endarterectomy or carotid artery stenting
* Recent major stroke with permanent neurological deficit
* Recent myocardial infarction within the past 3 months
* History of traumatic brain injury within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing elective carotid endarterectomy (CEA) under regional anesthesia at a single tertiary academic hospital. All participants must be able to tolerate awake surgery with regional anesthesia (superficial cervical plexus block) and undergo bilateral near-infrared spectroscopy (NIRS) monitoring and carotid stump pressure measurement during the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Carotid Stump Pressure Between Interhemispheric rSO₂ Symmetry and Asymmetry Groups | 3 minutes after carotid cross-clamping (intraoperative period)
  The primary outcome is the comparison of intraoperative carotid stump pressure (SP) between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂ difference) and those with nonsignificant asymmetry (≤10%).

SECONDARY OUTCOMES:
Interhemispheric asymmetry difference | 3 minutes after carotid cross-clamping (intraoperative period)
  This outcome is the absolute difference in percentage change (ΔrSO₂) between the ipsilateral (surgical) and contralateral hemispheres during carotid cross-clamping, measured using near-infrared spectroscopy (NIRS).
  Interhemispheric asymmetry is defined as:
  ΔrSO₂ = (Post-clamp rSO₂ - Pre-clamp rSO₂) / Pre-clamp rSO₂ × 100 Interhemispheric asymmetry difference = ΔrSO₂ Ipsilateral - ΔrSO₂ Contralateral
Correlation Between Carotid Stump Pressure and Interhemispheric ΔrSO₂ Difference | 3 minutes after carotid cross-clamping (intraoperative period)
  This outcome evaluates the relationship between carotid stump pressure and the absolute ΔrSO₂ difference between hemispheres (interhemispheric asymmetry) during carotid cross-clamping. The analysis will determine whether lower stump pressure values are significantly associated with increased interhemispheric cerebral oxygenation asymmetry.
Correlation Between Carotid Stump Pressure and Ipsilateral ΔrSO₂ | 3 minutes after carotid cross-clamping (intraoperative period)
  This outcome examines the association between carotid stump pressure and the percentage change in regional cerebral oxygen saturation (ΔrSO₂) specifically on the ipsilateral (surgical) hemisphere. ΔrSO₂ is calculated as the relative change from pre-clamp to post-clamp values using near-infrared spectroscopy (NIRS). The aim is to determine whether lower stump pressures are associated with greater ipsilateral desaturation, indicating impaired cerebral perfusion.
Carotid Stump Pressure Threshold Predictive of rSO₂ Asymmetry Using ROC Curve Analysis | 3 minutes after carotid cross-clamping (intraoperative period)
  This outcome evaluates whether a specific carotid stump pressure threshold can predict significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂ difference). Receiver operating characteristic (ROC) curve analysis will be used to calculate sensitivity, specificity, and area under the curve (AUC) for predictive accuracy.
Independent Predictive Value of Carotid Stump Pressure for rSO₂ Asymmetry in Multivariable Logistic Regression | 3 minutes after carotid cross-clamping (intraoperative period)
  This outcome assesses whether carotid stump pressure independently predicts the presence of interhemispheric rSO₂ asymmetry (>10%) during carotid cross-clamping. Logistic regression models will be adjusted for age, sex, degree of carotid stenosis, PaO₂, SpO₂, and systolic arterial pressure (SAP).
Comparison of Intraoperative Arterial Pressures Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This outcome includes the comparison of intraoperative systolic arterial pressure (SAP), diastolic arterial pressure (DAP), and mean arterial pressure (MAP), each measured in millimeters of mercury (mmHg), between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%).
Comparison of Intraoperative Heart Rate Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This outcome compares intraoperative heart rate (HR), measured in beats per minute (bpm), between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%).
Comparison of Intraoperative Arterial Oxygen Pressure (PaO₂) Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This outcome compares intraoperative arterial oxygen pressure (PaO₂), measured in millimeters of mercury (mmHg), between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%).
Comparison of Intraoperative Peripheral Oxygen Saturation (SpO₂) Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This outcome compares intraoperative peripheral oxygen saturation (SpO₂), expressed as a percentage (%), between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%).
Comparison of Cross-Clamp Duration, Total Surgical Time, and Total Anesthesia Time Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This outcome includes the comparison of three intraoperative time metrics - carotid cross-clamp duration, total surgical time, and total anesthesia time - each measured in minutes, between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%).
Comparison of Intraoperative Shunt Requirement Between Asymmetry and Symmetry Groups | Intraoperative period (from anesthesia start to end of surgery)
  This binary outcome compares the frequency of intraoperative shunt placement (yes/no) between patients with significant interhemispheric cerebral oxygenation asymmetry (>10% ΔrSO₂) and those with nonsignificant asymmetry (≤10%). The aim is to assess whether cerebral oxygenation asymmetry is associated with an increased need for shunting during carotid surgery.
Incidence of Postoperative Complications Within 30 Days | From date of surgery through postoperative day 30
  This outcome evaluates the incidence of postoperative complications occurring within 30 days after carotid endarterectomy. Complications of interest include new-onset neurological deficits (stroke, transient ischemic attack), bleeding requiring intervention, wound hematoma, or other clinically significant adverse events. Data will be collected through postoperative clinical assessments, follow-up visits, and review of medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Salih Tüzen, M.D:, Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Izmir Katip Celebi University Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data necessary to support the study protocol, including de-identified individual participant data (IPD) related to intraoperative monitoring (e.g., stump pressure values, rSO₂ measurements, hemodynamic parameters), primary and secondary outcome measures, and 30-day postoperative follow-up results, will be made available upon reasonable request from qualified researchers for academic purposes, in accordance with institutional and ethical guidelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT07150260/Prot_SAP_000.pdf